CLINICAL TRIAL: NCT06774742
Title: Evaluation of the Effects of a Dietary Supplement Containing a Full Range of Hyaluronic Acids in Healthy Female Subjects With Dry Facial Skin and Lips
Brief Title: Evaluation of the Effects of an Oral Supplementation Containing Hyaluronic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TS Biotech - Shandong Tiansheng Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-A01613-44
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-01

CONDITIONS: Skin Quality; Lips Quality; Persistence of the Effect
Keywords: skin hydration; skin quality; anti-aging; lips hydration; lips volume

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be double-blind. The products will be dispensed according to the randomization list by a responsible designated person other than the Investigator. The randomization list will be masked to the Investigator during the whole study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAFS Supplementation (Experimental): Hyaluronic acid full spectrum daily supplementation
  Interventions: Dietary Supplement: HAFS Supplementation
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HAFS Supplementation — 1 capsule of HAFS per day
  Arms: HAFS Supplementation
Dietary Supplement: Placebo — 1 capsule of placebo per day
  Arms: Placebo

SUMMARY:
This is a single center, double-blind, randomized, placebo-controlled study, performed on two parallel groups.

A total of 130 adult female subjects meeting specific inclusion/exclusion criteria will be included in order to have 120 subjects who complete the study at Day 98/Week 14.

Subjects will be randomly assigned to either the FS-HA oral supplementation group (60 subjects) or the placebo group (60 subjects).

The subjects should agree to attend a total of five (5) visits as follows:

* a screening visit within 21 days prior to Day 1 (from Day -22 to Day -1);
* a baseline visit (Day 1);
* two (2) intermediate visits (Day 29 and Day 84);
* a follow-up and end-of- study visit on Day 98.

The primary objective of this study is to evaluate the effects of an oral supplementation containing a FS-HA on facial skin hydration after 3 months of use, compared with Placebo.

The Secondary Objective(s) will evaluate the effects of an oral supplementation containing a FS-HA compared with Placebo on:

* the hydration of the lips using corneometry;
* the skin quality of the face using dermatological assessments and biophysical measurements (TEWL and Mexametry);
* the quality/health and beauty of the lips using dermatological assessments and biophysical measurements (Mexametry);
* the volume of the lips using image analysis;
* to assess the persistence of the effects 2 weeks after discontinuation;
* to assess the subject perceived efficacy and acceptability (subject self-assessment);
* to evaluate the safety of the study products.

ELIGIBILITY:
Inclusion Criteria:

1. Subject having signed an Informed Consent Form (ICF) before any trial related activity is carried out;
2. Female subject;
3. Subject aged 40 to 70 years inclusive at the time of signing the ICF;
4. Subject with thin and dry lips;
5. Subject with dry skin measured on the cheeks (corneometry < 50);
6. Female subject of childbearing potential must use one of the reliable methods of contraception during the investigation and agree not to change it during the study;
7. Subject willing and able to follow all the study procedures and restrictions and complete the whole study phase;
8. Subject affiliated to a health social security system (according to French Law).

Exclusion Criteria:

1. Female subject who is pregnant or who is breast feeding;
2. Female subject of childbearing potential with positive urine pregnancy test at the study visit (Day 1);
3. Women with a BMI ≤ 17 or ≥ 32 kg/cm²;
4. Subject with any uncontrolled diseases such as diabetes, hypertension, hyperthyroidism or hypothyroidism;
5. Presenting or having a history of eating disorder (e.g. anorexia, food allergy) or gastro-intestinal malabsorption such as celiac disease, Crohn's disease, lactose intolerance;
6. Subject with an history of sleeve or bypass
7. Subject with current participation in any other interventional clinical study, based on interview of the subject;
8. Subject with known or suspected hypersensitivity to any component(s) of the investigational products or to any ingredients of the vehicles (i.e., excipients);
9. Subject with skin abnormalities (e.g., scars, excessive hair, tattooing) or any dermatosis (e.g., psoriasis, eczema, acne vulgaris) on the face which could interfere with the study;
10. Subject having applied any cosmetic product (care cream, lotion, body milk…) or drug on the face (except usual cleansing products) within one week before the study visit (Day 1);
11. Subject impossible to contact in case of emergency;
12. Subject who, in the opinion of the investigator, is unlikely to comply with the Clinical Study Protocol (e.g., alcoholism, drug dependency or psychotic state);
13. Subject who is in an exclusion period in the National Biomedical Research Register of the French Ministry of Health at randomization;
14. Subject who has been deprived of their freedom by administrative or legal decision, or who is under care of a guardian or legal guardianship, or subject hospitalized in a medical or social establishment for any reason.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Skin hydration | Change from baseline to 3 months
  Facial skin hydration (Corneometer)

SECONDARY OUTCOMES:
Lip hydration | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  Changes in lip hydration (Corneometer®)
Lip color | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  Changes in skin and lip color (Mexameter®)
Lip volume | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  Change from baseline in lip volume (LifeViz®)
Skin barrier function | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  The measurement of the TEWL gives an indication of the integrity of the barrier function of the stratum corneum.
  The TEWL will be measured on the face at each evaluation visit using a Vapometer SWL-2 (Delfin, technologies, Kuopio, Finland). This portable device contains moisture sensors in a closed chamber type probe. The conditions of a closed chamber are created by contact with the skin surface (surface of the chamber =1 cm²). The TEWL measurement is expressed in g/m²/h after a stabilization time of 10 to 20 seconds.
Dermatological assessment of skin face | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  Scoring system for the assessment of the skin face
  Skin dryness : 0= no dryness to 9= very dry skin Skin roughness : 0= no roughness to 9= severe roughness Skin evenness : 0= not even at all to 9= very even Skin suppleness : 0= not supple at all to 9= very supple skin Skin elasticity : 0= no elasticity at all to 9= maximal elasticity Skin firmness 0= no firm at all to 9= very firm Skin plumping 0= not plump at all to 9= very plump
Dermatological assessment of lips | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  At each evaluation visit, the lip qualities will be assessed by the Investigator/evaluator using the following 6-point scoring system from 0 to 5.
  Lips fullness 0= very thin to 5= very full Lips dryness 0= no dryness to 5= very dry lips Lips roughness 0= no roughness to 5= severe roughness
Self assessment questionnaire | From baseline to Day 29, Day 84 and Day 98 (2 weeks after supplementation end)
  1. Evaluation of the skin face : wrinkle, hydration, firmness, softness, radiance, plump (scores from 0 (not) to 3 (high))
  2. Evaluation of the lips : hydration, volume, fine lines, color, gloss (scores from 0 being mild and 10 very strong)
  3. Evaluation of hair quality : volume, growth, loss, strength, radiance (scores from 0 (not) to 3 (high))
  4. Evaluation of the nail quality : strength, radiance, frailty, growth (scores from 0 (not) to 3 (high))
  5. Joint health

CONTACTS AND LOCATIONS:
Locations (1):
- CPCAD Hôpital L'Archet 2, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michelotti A, Cestone E, De Ponti I, Pisati M, Sparta E, Tursi F. Oral intake of a new full-spectrum hyaluronan improves skin profilometry and ageing: a randomized, double-blind, placebo-controlled clinical trial. Eur J Dermatol. 2021 Dec 1;31(6):798-805. doi: 10.1684/ejd.2021.4176. PMID 34933842
- [Background] Hsu TF, Su ZR, Hsieh YH, Wang MF, Oe M, Matsuoka R, Masuda Y. Oral Hyaluronan Relieves Wrinkles and Improves Dry Skin: A 12-Week Double-Blinded, Placebo-Controlled Study. Nutrients. 2021 Jun 28;13(7):2220. doi: 10.3390/nu13072220. PMID 34203487
- [Background] Gollner I, Voss W, von Hehn U, Kammerer S. Ingestion of an Oral Hyaluronan Solution Improves Skin Hydration, Wrinkle Reduction, Elasticity, and Skin Roughness: Results of a Clinical Study. J Evid Based Complementary Altern Med. 2017 Oct;22(4):816-823. doi: 10.1177/2156587217743640. Epub 2017 Dec 4. PMID 29228816
- [Background] Linkov G, Wick E, Kallogjeri D, Chen CL, Branham GH. Perception of upper lip augmentation utilizing simulated photography. Arch Plast Surg. 2019 May;46(3):248-254. doi: 10.5999/aps.2018.01319. Epub 2019 May 15. PMID 31113187
- [Background] Stojanovic L, Majdic N. Effectiveness and safety of hyaluronic acid fillers used to enhance overall lip fullness: A systematic review of clinical studies. J Cosmet Dermatol. 2019 Apr;18(2):436-443. doi: 10.1111/jocd.12861. Epub 2019 Jan 12. PMID 30636365
- [Background] Day AJ, de la Motte CA. Hyaluronan cross-linking: a protective mechanism in inflammation? Trends Immunol. 2005 Dec;26(12):637-43. doi: 10.1016/j.it.2005.09.009. Epub 2005 Oct 7. PMID 16214414
- [Background] Stern R, Asari AA, Sugahara KN. Hyaluronan fragments: an information-rich system. Eur J Cell Biol. 2006 Aug;85(8):699-715. doi: 10.1016/j.ejcb.2006.05.009. Epub 2006 Jul 5. PMID 16822580
- [Background] Tavianatou AG, Caon I, Franchi M, Piperigkou Z, Galesso D, Karamanos NK. Hyaluronan: molecular size-dependent signaling and biological functions in inflammation and cancer. FEBS J. 2019 Aug;286(15):2883-2908. doi: 10.1111/febs.14777. Epub 2019 Feb 21. PMID 30724463
- [Background] Heldin P, Lin CY, Kolliopoulos C, Chen YH, Skandalis SS. Regulation of hyaluronan biosynthesis and clinical impact of excessive hyaluronan production. Matrix Biol. 2019 May;78-79:100-117. doi: 10.1016/j.matbio.2018.01.017. Epub 2018 Jan 31. PMID 29374576
- [Background] Abatangelo G, Vindigni V, Avruscio G, Pandis L, Brun P. Hyaluronic Acid: Redefining Its Role. Cells. 2020 Jul 21;9(7):1743. doi: 10.3390/cells9071743. PMID 32708202
- [Background] Stern R. Hyaluronan catabolism: a new metabolic pathway. Eur J Cell Biol. 2004 Aug;83(7):317-25. doi: 10.1078/0171-9335-00392. PMID 15503855
- [Background] Gao YR, Wang RP, Zhang L, Fan Y, Luan J, Liu Z, Yuan C. Oral administration of hyaluronic acid to improve skin conditions via a randomized double-blind clinical test. Skin Res Technol. 2023 Nov;29(11):e13531. doi: 10.1111/srt.13531. PMID 38009035